CLINICAL TRIAL: NCT00779298
Title: Effect of Commercial Rye Whole-Meal Bread on Postprandial Blood Glucose and Gastric Emptying in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Other Study IDs: Dnr 709/2004
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: rye whole-meal bread; white-wheat bread; gastric emptying rate; postprandial glucose response; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy subjects: Healthy subjects, without symptoms or a prior history of gastrointestinal disease, abdominal surgery or diabetes mellitus

SUMMARY:
Increased intake of dietary fibre and whole grains is related to reduced risk of developing diabetes. The term "whole grain" is often used for whole-meal products in which the structure of the cereal grain is destroyed in the flour containing the original dietary fiber, but also for cereal products in which a large proportion of whole cereal grains is intact. The aim of this study was to evaluate the effect of commercial rye whole-meal bread (RWMB) compared to white-wheat bread (WWB) on gastric emptying rate (GER), postprandial glucose response in healthy subjects.

DETAILED DESCRIPTION:
Ten healthy subjects, without symptoms or a prior history of gastrointestinal disease, abdominal surgery or diabetes mellitus, were assessed by using a blinded crossover trial. The subjects were examined regarding blood glucose levels and GER after ingestion of 150g WWB or RWMB on two different occasions after an overnight fast. GER was measured using a standardized real time ultrasonography. GER was calculated as a percentage change in antral cross sectional area 15 and 90 minutes after the finished meal with WWB and RWMB. Finger-prick capillary samples were collected before and 40, 60, and 90 min after the start of the meal to measure blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* without symptoms or a prior history of gastrointestinal disease, abdominal surgery or diabetes mellitus

Exclusion Criteria:

* with symptoms or prior history of gastrointestinal disease, abdominal surgery or diabetes mellitus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects were recruited from the population in a southern county of Sweden.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Medicine, Malmö University Hospital,, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Hlebowicz J, Jonsson JM, Lindstedt S, Bjorgell O, Darwich G, Almer LO. Effect of commercial rye whole-meal bread on postprandial blood glucose and gastric emptying in healthy subjects. Nutr J. 2009 Jun 16;8:26. doi: 10.1186/1475-2891-8-26. PMID 19531257